CLINICAL TRIAL: NCT06403306
Title: Comparative Evaluation of the Success of Er,Cr:YSGG Laser Pulpotomy With Ferric Sulfate and Ankaferd in Primary Molar Teeth
Brief Title: Evaluation of Pulpotomy Success of Different Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, NECIBE DAMLA ŞAHIN, Lecturer, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/08
Record Dates: First submitted 2024-04-27; First posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pulpal Bleeding; Staining; Primary Teeth; Pulpotomy
MeSH Terms: interventions — ferric sulfate; ankaferd blood stopper; Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ferric Sulfate (Active Comparator): Ferric Sulfate (FS), widely used in pulpotomy treatment of primary teeth, provides hemostasis through a chemical reaction with blood. The FS solution was kept in the cavity for 15 seconds using cotton pellets in the FS group.
  Interventions: Drug: Ferric Sulfate (Viskostat; Ultradent, Utah, USA)
- Ankaferd Blood Stopper (Experimental): Ankaferd Blood Stopper (ABS), recently introduced to clinical practice as an alternative to FS, is a herbal hemostatic agent. The ABS solution drawn from the 1 ml ampoule to the syringe according to the manufacturer's instructions, was kept in the cavity for 15 seconds using cotton pellets in the ABS group.
  Interventions: Drug: Ankaferd Blood Stopper (Ankaferd Blood Stopper, Ankaferd Ilaç Kozmetik A.S, Istanbul, Turkey)
- Er,Cr:YSGG laser (Experimental): Er,Cr:YSGG laser was applied in a non-contact manner on the pulp tissue from a distance of 3-4 mm for ten seconds, with an energy intensity of 25 mL, output power of 0.5 W, and frequency of 20 Hz. The MZ6 laser tip was used for application.
  Interventions: Device: Er,Cr:YSGG laser (Waterlase MD, Biolase, USA)

INTERVENTIONS:
Drug: Ferric Sulfate (Viskostat; Ultradent, Utah, USA) — Widely used in pulpotomy treatment of primary teeth, provides hemostasis through a chemical reaction with blood. The metal-protein complex, formed due to contact with blood, creates a mechanical plug; thus, hemostasis occurs without clot formation.
  Other Names: Viskostat
  Arms: Ferric Sulfate
Drug: Ankaferd Blood Stopper (Ankaferd Blood Stopper, Ankaferd Ilaç Kozmetik A.S, Istanbul, Turkey) — Recently introduced to clinical practice as an alternative to FS, is a herbal hemostatic agent. It consists of a standardized mixture of Thymus vulgaris (thyme), Alpinia officinarum (galangal), Vitis vinifera (vine), Glycyrrhiza glabra (licorice) and Urtica dioica (nettle).
  Other Names: not
  Arms: Ankaferd Blood Stopper
Device: Er,Cr:YSGG laser (Waterlase MD, Biolase, USA) — Alternative technique introduced to clinical practice in recent years to provide hemostasis in vital pulp treatment is the usage of lasers in various wavelengths. Using lasers in pulpotomy provides many advantages such as tissue vaporization and coagulation, maintenance of a blood-free working field due to its property to close small blood vessels, minimal clot formation, and sterilization of the wound surface. Furthermore, laser systems were reported to induce cellular biostimulation. Er,Cr:YSGG lasers which belong to the Erbium laser family are the laser systems with the highest absorption rate by water, having a wavelength of 2780 nm. Besides, Erbium lasers manifest bactericidal effects.
  Other Names: Waterlase
  Arms: Er,Cr:YSGG laser

SUMMARY:
Considering the lack of data in the literature concerning the success of Er,Cr:YSGG laser in pulpotomy treatment of primary teeth, the present study aimed to compare this laser system with two different chemical hemostatic agents regarding its clinical and radiographic success.

DETAILED DESCRIPTION:
The study was carried on 65 patients (33 females and 32 males) with ages ranging between 5-9 years and having no systemic disease. Inclusion criteria were as follows; deep dentin caries, lack of spontaneous pain, no sensitivity to percussion and palpation, no soft tissue pathologies such as edema, fistula, abscess, mechanical exposure greater than pinpoint, carious exposure, suitability for restoration with stainless steel crowns, healthy lamina dura and periodontal space, no radiographic pathologies in the interradicular and periapical regions, no pathological external and internal resorption, and no calcified masses within the pulp. Only the mandibular primary molars were included in the study to evaluate the roots better radiologically. A single physician performed all patients' treatments. Following administration of local anesthesia, the teeth were isolated by a rubber dam. The carious enamel tissue was removed and the cavities were formed using a high-speed rotary instrument under water cooling. The carious dentin was removed using a low-speed rotary instrument and steel round bur. In the teeth included in the study, after opening the access cavity, the coronal pulp was removed with a sharp, sterile excavator and low-speed rotary instrument, and the pulp chamber was rinsed with saline. Primary bleeding control was provided in all groups by applying moisturized sterile cotton pellets over the canal orifices for five minutes with minimal pressure. The teeth in which bleeding could not be controlled within five minutes were excluded from the study, and root canal treatment was performed in these teeth. In the teeth that bleeding control was provided, FS, ABS, or Er,Cr:YSGG laser applications were made according to the order on the randomization list.

Following the primary bleeding control, the FS solution was kept in the cavity for 15 seconds using cotton pellets in the FS group. The ABS solution drawn from the 1 ml ampoule to the syringe according to the manufacturer's instructions, was kept in the cavity for 15 seconds using cotton pellets in the ABS group. In the laser group, both the physician and the patient wore protective glasses before the procedure. Er,Cr:YSGG laser (Waterlase MD, Biolase, USA) was applied in a non-contact manner on the pulp tissue. In all groups, after secondary bleeding control, the pulp chamber was sealed with zinc oxide -eugenol (ZOE). Glass ionomer cement was applied over the ZOE base and teeth were restored with stainless steel crown. Following the treatment, the patients were called for follow-up examinations at intervals of 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* deep dentin caries, lack of spontaneous pain, no sensitivity to percussion and palpation
* no soft tissue pathologies such as edema, fistula, abscess
* mechanical exposure greater than pinpoint, carious exposure,
* suitability for restoration with stainless steel crowns
* healthy lamina dura and periodontal space, no radiographic pathologies in the interradicular and periapical regions, no pathological external and internal resorption, and no calcified masses within the pulp
* mandibular primary molar

Exclusion Criteria:

* maxiller primary molar
* teeth with radiographic pathology

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 81 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | Following the treatment, the patients were called for follow-up examinations at intervals of 3 months for 12 months.
  In clinical examination, treatment was considered unsuccessful when one of the following findings were detected: Spontaneous pain, tenderness to percussion and palpation, fistula formation, soft tissue swelling, and pathological mobility. In teeth in which treatment was considered unsuccessful, root canal treatment or extraction was performed according to the cause of the failure. When indicated, a space maintainer was applied following extraction.
Radiographic success rate | Following the treatment, the patients were called for follow-up examinations at intervals of 3 months for 12 months.
  In the radiological examination, presence of periapical and/or interradicular radiolucency, widening of the periodontal ligament, loss of lamina dura, the presence of internal or external pathological resorption were considered as failure. In teeth in which treatment was considered unsuccessful, root canal treatment or extraction was performed according to the cause of the failure. When indicated, a space maintainer was applied following extraction.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Arıkan, Study Director — Kırıkkale University
Locations (1):
- Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodd HD, Waterhouse PJ, Fuks AB, Fayle SA, Moffat MA; British Society of Paediatric Dentistry. Pulp therapy for primary molars. Int J Paediatr Dent. 2006 Sep;16 Suppl 1:15-23. doi: 10.1111/j.1365-263X.2006.00774.x. No abstract available. PMID 16939452
- [Background] Vargas KG, Packham B, Lowman D. Preliminary evaluation of sodium hypochlorite for pulpotomies in primary molars. Pediatr Dent. 2006 Nov-Dec;28(6):511-7. PMID 17249432
- [Background] Goker H, Haznedaroglu IC, Ercetin S, Kirazli S, Akman U, Ozturk Y, Firat HC. Haemostatic actions of the folkloric medicinal plant extract Ankaferd Blood Stopper. J Int Med Res. 2008 Jan-Feb;36(1):163-70. doi: 10.1177/147323000803600121. PMID 18304416
- [Background] Chandran V, Ramanarayanan V, Menon M, Varma B, Sanjeevan V. Effect of LASER therapy Vs conventional techniques on clinical and radiographic outcomes of deciduous molar pulpotomy: A systematic review and meta-analysis. J Clin Exp Dent. 2020 Jun 1;12(6):e588-e596. doi: 10.4317/jced.56436. eCollection 2020 Jun. PMID 32665819
- [Background] Cengiz E, Yilmaz HG. Efficacy of Erbium, Chromium-doped:Yttrium, Scandium, Gallium, and Garnet Laser Irradiation Combined with Resin-based Tricalcium Silicate and Calcium Hydroxide on Direct Pulp Capping: A Randomized Clinical Trial. J Endod. 2016 Mar;42(3):351-5. doi: 10.1016/j.joen.2015.11.015. Epub 2015 Dec 23. PMID 26723484
- [Background] Betancourt P, Merlos A, Sierra JM, Camps-Font O, Arnabat-Dominguez J, Vinas M. Effectiveness of low concentration of sodium hypochlorite activated by Er,Cr:YSGG laser against Enterococcus faecalis biofilm. Lasers Med Sci. 2019 Mar;34(2):247-254. doi: 10.1007/s10103-018-2578-6. Epub 2018 Jul 6. PMID 29980946
- [Background] Fahim SZ, Ghali RM, Hashem AA, Farid MM. The efficacy of 2780 nm Er,Cr;YSGG and 940 nm Diode Laser in root canal disinfection: A randomized clinical trial. Clin Oral Investig. 2024 Feb 26;28(3):175. doi: 10.1007/s00784-024-05563-z. PMID 38403667